CLINICAL TRIAL: NCT05816408
Title: Effect of Breast Milk Feeding on Critically Ill Neonates
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mohsen Ezzat, Principal Investigator, Assiut University
Other Study IDs: Effect of breast milk feeding
Record Dates: First submitted 2023-03-17; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Globally, the estimated preterm birth rate is estimated at 10.6% of all live births, or about 14.8 million infants per year. Breastfeeding is associated with a reduction of risk for several acute and chronic diseases in women and their infants, and the benefits are especially important for small, sick and preterm infants. Important benefits of breastmilk provision for premature and fragile infants including a reduction of the risk for late-onset sepsis, necrotizing enterocolitis, and ventilator-associated pneumonia.

In 2020, the World Health Organization (WHO) and the United Nations Children's Fund (UNICEF) released The Baby friendly Hospital Initiative (BFHI) for small, sick and preterm newborns. Based on the evidence put forward in this document,this review outlines the main steps that health care professionals and facilities can take to support breastfeeding in vulnerable groups of infants. The objective of this study is to summarize essential steps for healthcare personnel and health care facilities to improve breastfeeding practices in small, sick and preterm infants.

DETAILED DESCRIPTION:
Globally, the estimated preterm birth rate is estimated at 10.6% of all live births, or about 14.8 million infants per year. Breastfeeding is associated with a reduction of risk for several acute and chronic diseases in women and their infants, and the benefits are especially important for small, sick and preterm infants. Important benefits of breastmilk provision for premature and fragile infants including a reduction of the risk for late-onset sepsis, necrotizing enterocolitis, and ventilator-associated pneumonia.

In 2020, the World Health Organization (WHO) and the United Nations Children's Fund (UNICEF) released The Baby friendly Hospital Initiative (BFHI) for small, sick and preterm newborns. Based on the evidence put forward in this document,this review outlines the main steps that health care professionals and facilities can take to support breastfeeding in vulnerable groups of infants. The objective of this study is to summarize essential steps for healthcare personnel and health care facilities to improve breastfeeding practices in small, sick and preterm infants.

Breastfeeding initiation and skin-to-skin care Providers should support all mothers and infants with immediate skin-to-skin care (SSC) after birth and assist mothers to initiate breastfeeding (or breastmilk expression and feedings) as soon as possible. A systematic review and meta-analysis on very early breastfeeding initiation and neonatal mortality in 136,047 infants found that breastfeeding initiation 2_23 h after birth was associated with a 33% higher risk of mortality compared to breastfeeding initiation _1 h after birth, however potential confounding by factors such as health challenges causing both delayed initiation and increased mortality needs to be considered.

Skin-to-skin care improves breastfeeding rates in very preterm infants. In infants with low-birth weight, evidence from a Cochrane review supports the use of skin to skin care for reduction of both infant mortality and morbidity, especially in low income settings.

Skin-to-skin care helps to stabilize infants' body temperature and blood sugar and helps to reduce infant procedural pain, even in very preterm neonates.It also stabilizes preterm infants' respiratory function, which isthought to be guided by the caregiver's cardiac rhythm. Compared to incubator care, cerebral oxygenation and other physiological parameters in ventilated preterm infants has not been shown to become more unstable during SSC with their mothers.Skin-to-skin contact has positive effects on the neonate's microbiome through population of the neonate's skin with beneficial bacteria and has been shown to decrease the risk of nosocomial infections. Regular and prolonged SSC can reduce the risk of hospital-acquired infections, bronchopulmonary dysplasia and cholestasis in a dose-dependent fashion, even in very preterm infants.

Responsive (on-demand) breastfeeding means following an infant's feeding cues to guide feeding times. If the infant does not have contraindications to enteral feeding, breastfeeding or feeding of expressed human milk can be initiated as soon as the infant has stable vital signs, which most of the time can begin within the first few hours of life.Because preterm infants are neurologically immature, responsive feeding may not be possible initially. However,as preterm infants mature, semi-demand feeding can be started, which means that breastfeeding is initiated in response to infant cues, but ended when the infant stops suckling.

Exclusive breastfeeding rates for premature infants have been shown to drop significantly after discharge. Healthcare teams can support families through connecting them to clinical and community-based referrals after hospital discharge (e.g. paediatricians , lactation consultants, breastfeeding peer support groups). Beyond referrals, healthcare professionals should bear in mind that the hospitalization period for small, sick or preterm neonates may pose challenges to bonding and attachment and parents' confidence as caregivers. Therefore, preparing parents for bringing fragile infants home is essential.Qualitative studies with parents of neonates have demonstrated that parents value dialogue and timely communication with the healthcare team prior to discharge. These studies underline the importance of including support persons (fathers or partners) in conversations and planning for the transition home.Preterm infants exclusively breastfed after discharge are at increased risk of low lean body mass and low bone mineral density, and continued provision of fortifier in addition to breastfeeding after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with critical illness as RDS,pneumonias,perinatal asphyxia,enterocolitis,meconium aspiration syndrome,neonatal sepsis diagnosed on the basis of clinical signs and symptoms

Exclusion Criteria:

* neonates cannot breastfeed due to GIT anomalies as esophageal atresia, duodenal atreaia ,congenital hypertrophic pyloric stenosis , intestinal obstruction , metabolic diseases ,complex cardic anomalies

Max Age: 28 Days | Sex: All
Age Groups: Child
Study Population: 50 neonates aged (0-28 days)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of critically ill neonates who receiving breast milk and affect on their weight gain | Baseline
  This study was aimed to assess the effect of breast milk feeding on critically ill neonates regarding weight gain.
Number of critically ill neonates who receiving breast milk and affect on their reflexes | Baseline
  This study was aimed to assess the effect of breast milk feeding on critically ill neonates regarding reflexes.
Number of critically ill neonates who receiving breast milk and affect on their starting of enteral feeding | Baseline
  This study was aimed to assess the effect of breast milk feeding on critically ill neonates regarding start of enteral feeding
Number of critically ill neonates who receiving breast milk and affect on their durtation to stay on mechanical ventilation | Baseline
  This study was aimed to assess the effect of breast milk feeding on critically ill neonates regarding the stay on mechanical ventilation.
Number of critically ill neonates who receiving breast milk and affect on their duration of hospital stay | Baseline
  This study was aimed to assess the effect of breast milk feeding on critically ill neonates regarding duration of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Salah El-Din Amry, Prof, Principal Investigator — Assiut University; Amira Mohamed, Assist prof, Principal Investigator — Assiut University